CLINICAL TRIAL: NCT01128088
Title: The Stress Response in Laparoscopic Colorectal Surgery and Its Role in the Development of the Enhanced Recovery Program.
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: SURGN0008
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Laparoscopy; Colorectal Disease; Stress Response
Keywords: Enhanced recovery program in laparoscopic surgery
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- PCA and Volulyte
- PCA and Hartmann's
- Spinal and Volulyte
- Spinal and Hartmann's

SUMMARY:
Keyhole bowel surgery provides the patient with an improved outcome following surgery in comparison to more traditional surgery requiring a large cut. In order to further improve outcomes there are several variables that must be controlled before, during and after the operation. These variables are the correct pain relief, accurate control and measurement of the fluid that is given during the operation and the subsequent mobility following surgery. Previous research has already identified that an enhanced recovery program (careful control and structure to the patients journey) will reduce the length of stay and complications after an operation. Currently an integral part of the enhanced recovery program requires the use of an epidural (a thin tube in the spine) to provide continuous pain relief for up to 48 hours. Through research previously undertaken at the MATTU the investigators have shown that an epidural can lead to an increase in the length of stay and a delay in the return to normal bowel function. A reason for the use of an epidural is to suppress the stress response.

The investigators aim to recruit patients from outpatient clinic undergoing keyhole bowel surgery in one unit and randomize them to receive one of two different pain relief methods after the operation. Patients will follow the same care as standard patients but their pain relief will differ between two already well established modalities. They will also receive different intravenous fluids. Blood will also be drawn at various intervals immediately after the operation for future analysis. The trial will be funded by the MATTU and will run for approximately 18 months. This trial will enable us to establish the stress response in the four groups and correlate it to the patient's outcome with an aim to refining the enhanced recovery program.

ELIGIBILITY:
Inclusion Criteria:

* Colonic or rectal resection procedure.

Exclusion Criteria:

* Stoma formation (previous research at the MATTU has shown that the formation of a stoma significantly affects the quality of life to the degree that there is no difference between open and laparoscopic surgery)

  * Conversion to a traditional open operation (removes the elements of keyhole surgery)
  * Contraindication to spinal anaesthesia: abnormal clotting, skin infection over or near the back, presence of neurological disorders or anatomical abnormalities of the vertebral column. (For patient safety)
  * Contraindication to the use of oesophageal Doppler: oesophageal disease, recent oesophageal surgery or upper airway surgery, moderate to severe aortic valve disease and any condition that causes bleeding problems. (For patient safety)
  * Diagnosis of diabetes mellitus (will confound the stress response analysis)
  * Treatment with exogenous steroids in the proceeding 3 months (will confound the stress response analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having colorectal resections at The Royal Surrey County Hospital
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The change in interleukin 6 levels following surgery for the four groups. | Change detected between 0 and 6 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Tim Rockall, MBBS FRCS MD, Study Director — Minimal Access Therapy Training Unit
Locations (1):
- The Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Day AR, Smith RV, Scott MJ, Fawcett WJ, Rockall TA. Randomized clinical trial investigating the stress response from two different methods of analgesia after laparoscopic colorectal surgery. Br J Surg. 2015 Nov;102(12):1473-9. doi: 10.1002/bjs.9936. Epub 2015 Sep 23. PMID 26395762